CLINICAL TRIAL: NCT06007521
Title: Validation of a Clinical Assessment Scale Specific to Alternating Hemiplegia
Acronym: TREAT-AHC
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0804
Record Dates: First submitted 2023-08-08; First posted 2023-08-23 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Alternating Hemiplegia
Keywords: Alternating Hemiplegia of Childhood; rating scale
MeSH Terms: conditions — Alternating hemiplegia of childhood | interventions — Interviews as Topic; Neurologists

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with alternating hemiplegia: Patients with alternating hemiplegia, from 0 to 99 years old
  Interventions: Other: interview with neurologist

INTERVENTIONS:
Other: interview with neurologist — interview with neurologist

SUMMARY:
Alternating Hemiplegia of Childhood (AHC) is a very rare neurological disorder of genetic origin, combining paroxysmal episodes and neurodevelopmental impairment. The disease is generally sporadic, and its incidence has been estimated at 1 in 100,000 births, with around 500 cases published worldwide. The true prevalence of AHC may be underestimated due to a lack of understanding of the disease and a high degree of phenotypic heterogeneity.

It should be noted that, to date, it is difficult to assess the clinical characteristics of AHC patients in a homogeneous way. The lack of disease-specific clinical outcome measures therefore constitutes a critical node for advancing AHC research. In addition, recognition of the pattern of movement disorders and the ability to classify their severity are very important and useful for the clinician. Homogeneous disease assessment will help plan rehabilitative and pharmacological interventions, facilitate monitoring of treatment outcomes, and predict prognosis.

This is why an AHC assessment scale have been developed in collaboration with clinical teams from the IAHCRC consortium.

The scale has already been tested and validated on Italian and Spanish patients. The aim of this study is therefore to validate the use of this same scale on our French population of AHC patients. The hypothesis of the study is that the practical use of this scale specific to alternating hemiplegia is reproducible. To this end, all the items on the scale will be scored independently for each patient by 4 neuropediatricians with expertise in the disease, in order to observe the reproducibility of the results obtained with this scale. The scale will be used for twenty AHC patients of all ages.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed diagnosis of AHC, unrestricted age range 0-99 years
* At least one parent and/or legal guardian who understands and speaks the national language

Adult patients :

* Gathering of the non-opposition of the patient and/or his legal representative

Minor patients :

* Collection of non-opposition from parents/guardians

Exclusion Criteria:

* Patient's refusal to participate in the study
* Patient under court protection, unable to give consent

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients likely to participate in the study will be identified within the ESEFNP Department - Clinical Epileptology, Sleep Disorders, Functional Child Neurology, Hôpital Femme Mère Enfant, (HCL) as part of their regular medical follow-up. 20 AHC patients will be included in this study.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2023-11-18 (Actual); Primary Completion 2023-11-19 (Actual); Study Completion 2023-11-19 (Actual)

PRIMARY OUTCOMES:
Composite primary endpoint : - missing data from the scale <5 - mean scores compared between the 4 neurologists are close to the scale's mid-point, i.e. floor and ceiling effects are < 20%, and skewness statistics are between 21 and 11 | At inclusion
  All statistical tests will be performed using SPSS version 24.0 statistical software, and P < 0.05 will be considered significant.
  Validation of the use of the scale based on the results obtained independently by the 4 expert neurologists using a composite primary endpoint consisting of three criteria:
  * missing data from the scale <5
  * mean scores compared between the 4 neurologists are close to the scale's mid-point, i.e. floor and ceiling effects are < 20%, and skewness statistics are between 21 and 11.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Epileptologie Clinique, des Troubles du Sommeil et de Neurologie Fonctionnelle de l'Enfant, Bron, Rhone, France

IPD SHARING:
Plan to Share IPD: No